CLINICAL TRIAL: NCT07003061
Title: The Effects of Sarcopenia on Neuromuscular Block in Gastrointestinal Cancer Surgery
Brief Title: Sarcopenia and Neuromuscular Block in Gastrointestinal Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Kemal ŞAHİN, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-05/79
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Cancer; Sarcopenia; Neuromuscular Blockade
MeSH Terms: conditions — Gastrointestinal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenic: Patients with gastrointestinal cancer scheduled for elective surgery who are identified as sarcopenic based on preoperative abdominal CT scans at the L3 vertebral level, according to established cut-off values.
  Interventions: Procedure: Standard Anesthesia Management
- Non-Sarcopenic: Patients with gastrointestinal cancer scheduled for elective surgery who are identified as non-sarcopenic based on preoperative abdominal CT scans at the L3 vertebral level, according to established cut-off values.
  Interventions: Procedure: Standard Anesthesia Management

INTERVENTIONS:
Procedure: Standard Anesthesia Management — All patients will receive standard anesthesia care as per institutional protocols. No experimental intervention will be applied.

SUMMARY:
This prospective observational study aims to evaluate the effects of sarcopenia on intraoperative neuromuscular block (NMB) in patients undergoing gastrointestinal cancer surgery. Adult patients scheduled for elective gastrointestinal cancer surgery will be grouped as sarcopenic or non-sarcopenic based on preoperative abdominal CT scans. Neuromuscular block parameters, including onset time, depth, duration, and recovery, will be objectively measured using TOF (Train-of-Four) monitoring. The study seeks to determine whether sarcopenia influences sensitivity to muscle relaxants and to contribute to individualized anesthesia management and patient safety.

DETAILED DESCRIPTION:
Sarcopenia, characterized by the loss of skeletal muscle mass and function, is a significant clinical parameter affecting both prognosis and perioperative management in patients with gastrointestinal (GI) cancer. It may alter the pharmacokinetic and pharmacodynamic properties of anesthetic agents, particularly neuromuscular blocking agents. This prospective observational study will be conducted at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital between June 1, 2025, and September 1, 2025.

Adult patients (aged 18 and above) scheduled for elective GI cancer surgery who have undergone preoperative abdominal computed tomography (CT) will be included. Patients with neuromuscular diseases, those on chronic steroid or immunosuppressive therapy, or those with significant organ failure will be excluded. Preoperative CT images at the L3 vertebral level will be evaluated by a radiologist to determine sarcopenia status, and patients will be divided into sarcopenic and non-sarcopenic groups according to established cut-off values.

All patients will receive standard anesthesia monitoring, including TOF (Train-of-Four) neuromuscular monitoring. The study will not alter any treatment protocols. After administration of muscle relaxants during anesthesia induction, neuromuscular block parameters such as onset time, depth, duration, need for reversal agents, and recovery time will be recorded. Demographic data, comorbidities, laboratory findings, type of surgery, and details of muscle relaxant use will also be collected.

The primary objective is to compare intraoperative neuromuscular block parameters between sarcopenic and non-sarcopenic patients. Statistical analysis will be performed using appropriate parametric or non-parametric tests for continuous variables and chi-square tests for categorical variables. The study aims to provide evidence for individualized dosing of muscle relaxants and to improve patient safety in anesthesia practice for GI cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients diagnosed with gastrointestinal system (GIS) cancer and scheduled for elective surgery
* Patients who have undergone preoperative abdominal computed tomography (CT) imaging
* Patients classified as American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Patients with a history of neuromuscular diseases
* Patients receiving chronic steroid or immunosuppressive therapy
* Patients with electrolyte imbalance
* Patients using medications that affect neuromuscular transmission
* Patients with severe organ failure in the preoperative period (e.g., liver or renal failure)
* Patients who refuse to participate in the study
* Patients requiring emergency surgery
* Patients using muscle relaxants in the preoperative period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 75 years who have been diagnosed with gastrointestinal cancer and are scheduled for elective surgery at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. All participants will have undergone preoperative abdominal CT scans. Both male and female patients meeting the inclusion and exclusion criteria will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Onset Time of Neuromuscular Block | Intraoperative (from induction until adequate block is achieved)
  Time from administration of the muscle relaxant to achievement of adequate neuromuscular block, measured by Train-of-Four (TOF) monitoring.
Depth of Neuromuscular Block (TOF Ratio) | Intraoperative (from induction to end of surgery)
  Intraoperative depth of neuromuscular block, continuously monitored using TOF ratio.
Duration of Neuromuscular Block | Intraoperative (from muscle relaxant administration to recovery)
  Time from administration of the muscle relaxant to recovery of neuromuscular function (TOF ratio ≥ 0.9).
Dose and Duration of Reversal Agent | Intraoperative (from administration of reversal agent to recovery)
  Total dose and time required for the reversal agent to achieve recovery from neuromuscular block.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal SAHIN, Principal Investigator — Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation; Mensure KAYA, Principal Investigator — Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation; Belkis YILMAZ, Principal Investigator — Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation; Ahmet BAYRAK, Principal Investigator — Ankara Oncology Education and Research Hospital Clinic of Radiology
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Rea, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will be made available upon reasonable request after publication of the study results.

REFERENCES:
- [Background] Almeida PS, Barao K, Forones NM. SARCOPENIA AND GASTROINTESTINAL CANCER: NUTRITIONAL APPROACH FOCUSING ON CURCUMIN SUPPLEMENTATION. Arq Gastroenterol. 2025 Apr 4;62:e24068. doi: 10.1590/S0004-2803.24612024-068. eCollection 2025. PMID 40197883
- [Background] Clark BC. Neuromuscular Changes with Aging and Sarcopenia. J Frailty Aging. 2019;8(1):7-9. doi: 10.14283/jfa.2018.35. PMID 30734824